CLINICAL TRIAL: NCT01543048
Title: Prognostic Value of Human Papillomavirus (HPV) Detection in Cervical Intra-epithelial Neoplasia (CIN) Recurrence After Conization: Prospective Study With Virological Follow-up on 24 Months (SUIVICOL)
Brief Title: Prognostic Value of Human Papillomavirus (HPV) Detection in Cervical Intra-epithelial Neoplasia (CIN) Recurrence After Conization
Acronym: SUIVICOL
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2010/18
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: CIN2/3 Recurrence
Keywords: Human Papilloma Virus (HPV); Virological tests; CIN3; Cervical cancer; Conization; within women treated by conization for a CIN3
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Follow-Up Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with CIN3 treated by conization
  Interventions: Other: Study Follow-Up

INTERVENTIONS:
Other: Study Follow-Up — Colposcopy (+/- biopsies), cytology, and virology tests will be performed at the time of conization and during the follow-up period (6, 12, 24 months). HPV expression will be assessed by centralized validated marketed tests (Hybrid Capture 2, RLA genotyping, PreTect® HPV-Proofer) and by a real time PCR measuring E2, E6 and E7 viral load of HPV 1.

SUMMARY:
CIN2/3 have been increased for many years and mainly concern women aged 25-29 years. They are subsequent to a persistent HPV infection and are classically treated by conization. Recurrences occur in 7 to 18 % of cases, mainly after CIN3 management during the first 2 years of follow-up. Follow-up is crucial to detect and treat recurrence and to select high risk women who might develop cervical cancer. Colposcopy and cytology have been recommended since 1989 by French ANAES, but these methods have poor sensitivity and specificity. However, DNA HPV testing is more sensitive and has demonstrated a very high negative predictive value, while specificity and positive predictive value remain average. Other HPV markers like genotyping, viral load and integration begin to be used in screening but have not been investigated in CIN2/3 follow-up to assess the values of various HPV markers which predict CIN2/3 recurrence after conization. The primary objective is to describe HPV expression (genotyping, viral load, mRNA E6 and E7) at the time of conization and during the follow-up period (6, 12, 24 months) and to assess the prognostic value of HPV 16 expression (viral load, mRNA E6 and E7) to determine the risk of CIN2/3 recurrence after conization, compared to the other clinical and virological risk factors.

DETAILED DESCRIPTION:
Women with CIN3 treated by conization will be consecutively included in this study during 12 months. They will be recruited in the 3 main University Hospitals of South West France (Bordeaux, Toulouse, Limoges) and followed-up for 24 months. Colposcopy (+/- biopsies), cytology, and virology tests will be performed at the time of conization and during the follow-up period (6, 12, 24 months). HPV expression will be assessed by centralized validated marketed tests (Hybrid Capture 2, RLA genotyping, PreTect® HPV-Proofer) and by a real time PCR measuring E2, E6 and E7 viral load of HPV 1.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years
* CIN 2 or 3 diagnosis at inclusion confirmed for a CIN3 diagnosis by conization.
* HPV detected by Hybrid Capture 2 or RLA genotyping.
* Informed and signed consent by the patient and the investigator
* Coverage by French social security

Exclusion Criteria:

* Pregnancy at the time of inclusion.
* Previous history conization.
* Atypical endometrial or glandular cells or evidence of carcinoma on conization.
* Previous vaccination with a prophylactic HPV vaccine.
* Active viral infections including HIV.
* Acquired or congenital immunodeficiency.
* Long term treatment by corticosteroids or immunosuppressive drugs.
* Persons under protection of law.
* Patients unable to meet the requirements of the protocol.
* Any condition that, according to the investigator, would prevent participation in the study or interfere with the objectives of the study (refusal of supervision at the University Hospital, expected change of address within 3 years, etc)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with CIN3 treated by conization
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2012-03-06 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Recurrence of CIN2/3 diagnosed on colposcopy-directed biopsy | For each patient, 24 month after inclusion
  Biopsies will be carried out in cases of abnormal findings by colposcopy, cytological anomalies (ASC-US, ASC-H, LSIL, HSIL, cancer), and/or colpo-cytological discordance. The prognostic impact of HPV16 compared to the other HR-HPV on the recurrence of CIN2/3 will be assessed

SECONDARY OUTCOMES:
Evaluation of CIN2/3 diagnosis tests | For each patient, 24 month after inclusion
  Sensitivity, specificity, positive and negative predictive values of the following tests in the diagnosis of CIN2/3 after conization:
  * Cytology (at the ASC-US threshold)
  * Colposcopy (at the grade 2 abnormal transformation threshold)
  * Hybrid Capture 2 (positivity threshold: 2 pg/ml)
  * RLA genotyping (presence or not of HPV 16 and/or other HR-HPV)
  * PreTect® HPV-Proofer (presence or not of mRNA E6 and E7 of HPV 16, 18, 31, 33, 45)

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève CHÊNE, MD-PhD, Study Chair — USMR - University Hospital Bordeaux, France
Locations (4):
- France (4):
  - CHU de Bordeaux, Bordeaux
  - CHU de Limoges, Hôpital Mère Enfant, Limoges
  - CHU de Toulouse, Hôpital Paule de Viguier, Toulouse
  - CHU de Toulouse, Hôpital Rangueil, Toulouse